CLINICAL TRIAL: NCT02842411
Title: Risk Factors for Inadequate Bowel Preparation in Patients With Chronic Constipation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: 20160616-5
Record Dates: First submitted 2016-06-25; First posted 2016-07-22 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-08

CONDITIONS: Constipation
Keywords: bowel preparation; chronic constipation; risk factor
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- chronic constipation: patients with chronic constipation based on Rome Ⅳ

SUMMARY:
Chronic constipation is one of the risk factors of inadequate bowel preparation, which could influence the effect of colonoscopy. The risk factors associated with inadequate bowel preparation in constipated patients remains unclear. Here the investigators investigated the high risk factors which might have influence on bowel preparation quality in a prospective cohort of patients with functional constipation.

ELIGIBILITY:
Inclusion Criteria:

* 18-90
* Patients undergoing colonoscopy;
* Patients meeting the criteria of chronic constipation of Rome Ⅳ;

Exclusion Criteria:

* history of colorectal surgery;
* known of suspected colonic stricture or obstructing tumour;
* ulcerative colitis;
* Crohn's disease;
* irritable bowel syndrome;
* toxic colitis or megacolon;
* known or suspected bowel obstruction or perforation;
* pregnancy or lactation;
* unable to give informed consent;
* haemodynamically unstable.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients >=18 years old undergoing colonoscopy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
adequate rate of bowel preparation ≥6 with each segment ≥2 | 6 months
  The adequacy of bowel preparation is defined as Boston Bowel Preparation Scale (BBPS), a 4-point scoring system applied to each of 3 broad regions of the colon: the right side, the transverse section, and the left side. They were summed to give the total BBPS score, which ranged from 0 to 9.

SECONDARY OUTCOMES:
polyp detection rate | 6 months
insertion time | 6 months
withdrawal time | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, MD, Principal Investigator — Xijing Hospital of Digestive Disease; Mingxin Zhang, MD, Principal Investigator — Tang-Du Hospital; Shiyang Ma, MD, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University; Yujie Jing, MD, Principal Investigator — Chinese PLA 451 Hospital
Locations (4):
- China (4):
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - Chinese PLA 451 Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ness RM, Manam R, Hoen H, Chalasani N. Predictors of inadequate bowel preparation for colonoscopy. Am J Gastroenterol. 2001 Jun;96(6):1797-802. doi: 10.1111/j.1572-0241.2001.03874.x. PMID 11419832
- [Background] Hassan C, Fuccio L, Bruno M, Pagano N, Spada C, Carrara S, Giordanino C, Rondonotti E, Curcio G, Dulbecco P, Fabbri C, Della Casa D, Maiero S, Simone A, Iacopini F, Feliciangeli G, Manes G, Rinaldi A, Zullo A, Rogai F, Repici A. A predictive model identifies patients most likely to have inadequate bowel preparation for colonoscopy. Clin Gastroenterol Hepatol. 2012 May;10(5):501-6. doi: 10.1016/j.cgh.2011.12.037. Epub 2012 Jan 10. PMID 22239959
- [Result] Suares NC, Ford AC. Prevalence of, and risk factors for, chronic idiopathic constipation in the community: systematic review and meta-analysis. Am J Gastroenterol. 2011 Sep;106(9):1582-91; quiz 1581, 1592. doi: 10.1038/ajg.2011.164. Epub 2011 May 24. PMID 21606976
- [Derived] Guo X, Shi X, Kang X, Luo H, Wang X, Jia H, Tao Q, Wang J, Zhang M, Wang J, Lu X, Ma S, Lin T, Jing Y, Pan Y, Guo X, Fan D. Risk Factors Associated with Inadequate Bowel Preparation in Patients with Functional Constipation. Dig Dis Sci. 2020 Apr;65(4):1082-1091. doi: 10.1007/s10620-019-05847-5. Epub 2019 Oct 12. PMID 31605278